CLINICAL TRIAL: NCT06485297
Title: Evaluation of the Tunnel Effect Within a French Population of Dental Surgeons: a Pilot Cross-sectional Study
Brief Title: Effect Tunnel in Oral Medicine
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Odonto02
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-09

CONDITIONS: Psychological
Keywords: tunnel effect

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Externs in 6th year: external in the 6th year working within the Riquier Institute of Oral Medicine at Nice University Hospital.
  Interventions: Other: questionnary
- Interns: interns working within the Riquier Institute of Oral Medicine at Nice University Hospital.
  Interventions: Other: questionnary
- Private practitioners: teachers working within the Riquier Institute of Oral Medicine at Nice University Hospital.
  Interventions: Other: questionnary
- CHU practitioners: several categories of dental surgeons, on the basis of a list of addresses provided by the school of the faculty of dental surgery of Côte d'Azur University
  Interventions: Other: questionnary

INTERVENTIONS:
Other: questionnary — questionnaire in word format, sent by email and in paper version, which was established by the two main investigators (Diana Neponoceno, Pr Sophie-Myriam Dridi)

SUMMARY:
Evaluate whether there are differences in knowledge between practitioners and students regarding the tunnel effect, to validate the benefit of teaching it in oral medicine. Main objective: to evaluate the state of knowledge relating to the tunnel effect concerning the performance of a surgical procedure, of a cohort of odontologists of different professional levels. Secondary objectives: evaluate the nature of the means they propose in order to counter the effects of this cognitive bias.

ELIGIBILITY:
Inclusion Criteria: - Externs in the 6th year, interns and teachers working within the Riquier Institute of Oral Medicine at Nice University Hospital, and private dental surgeons.

Exclusion Criteria: - dental student under 6th year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6th year students and interns + CHU and liberal practitioners
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the state of knowledge relating to the tunnel effect concerning the performance of a surgical procedure, of a cohort of odontologists of different professional levels. | At the inclusion
  Questionnaire: 6 items. Main objective: to evaluate the state of knowledge relating to the tunnel effect concerning the performance of a surgical procedure, of a cohort of odontologists of different professional levels. The responses were compared to each other, following interpretation of the relevant data by Diana Neponoceno. Discrepancies in responses or inconsistencies were supported by studies confirming or refuting the results

SECONDARY OUTCOMES:
Evaluation of the nature of the means proposed to combat the tunnel effect | At the inclusion
  Secondary objectives: evaluate the nature of the means they propose in order to counter the effects of this cognitive bias. The responses were compared to each other, following interpretation of the relevant data by Diana Neponoceno. Discrepancies in responses or inconsistencies were supported by studies confirming or refuting the results

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France